CLINICAL TRIAL: NCT00917345
Title: Diagnosis of Primary Aldosteronism: Comparison of Post Captopril Active Renin Concentration and Plasma Renin Activity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Novartis (Industry)
Responsible Party: Yang PC, National Taiwan University Hospital
Other Study IDs: 200904076R
Record Dates: First submitted 2009-06-08; First posted 2009-06-10 (Estimated); Last update posted 2009-06-10 (Estimated); Status verified 2009-06

CONDITIONS: Primary Aldosteronism
Keywords: ARC; PRA; primary aldosteronism; captopril test; aldosterone-renin ratio; Primary aldosteronism (PA) than PRA and establish thresholds for the diagnosis using ARC.
MeSH Terms: conditions — Hyperaldosteronism; AIDS-Related Complex

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- aldosteronism, hypertension
  Interventions: Drug: captopril test
- hypertension
  Interventions: Drug: captopril test

INTERVENTIONS:
Drug: captopril test — The blood samplings were obtained one hour after the administration of 50 mg of captopril.The testing is performed in the morning on a seated ambulatory patient

SUMMARY:
Background: The most common pharmacologic test for diagnosis of primary aldosteronism (PA) is administration of captopril to examine whether abnormal aldosterone to plasma rennin activity (PRA)(ARR) persists, although active rennin concentration (ARC) in contrast to PRA may offers advantages with regard to processing and standardization.

Objective: To assess whether post captopril ARC offer any additional advantage in screening primary aldosteronism (PA) than PRA and establish thresholds for the diagnosis using ARC.

DETAILED DESCRIPTION:
Primary aldosteronism (PA), characterized by an inappropriate production of aldosterone, affects 5-13% of patients with hypertension(1, 2). The use of aldosterone-renin ratio (ARR) as screening test contributes to the increased diagnostic rate of this disease(2), but it is not standardized among laboratories. As the incidence of PA has increased since ARR has been used as a screening test (3, 4), the difficulty in establishing a diagnosis of PA may be encountered because of atypical manifestations. Administration of captopril to differentiate the normal renin-angiotensin- aldosterone axis from autonomous secretion of aldosterone has been proved to be a safe and effective test in confirmation of the diagnosis (5-8). Several studies have demonstrated that the ARR after a single dose of captopril is diagnostic (5-8) and as sensitive as the saline loading test for the identification of aldosterone- producing adenoma (APA)(8).

Active rennin concentration (ARC) is considerably easier to perform; being a single immunoradiometric assay as opposed to the initial generation of angiotensin I generated from angiotensinogen followed by radioimmunoassay of PRA(9). It was demonstrated as a reliable and convenient screening tool for ambulatory conditions, independent of body posture (10). Decreased angiotensinogen level is noted in pathological status ( e.g. liver cirrhosis, sever cardiac failure) (11, 12) that results in dissociate of PRA measurement. PAC when used in conjunction with aldosterone to produce an ARRARC , has been reported to classify aldosteronism correctly(13). Although PRA is highly sensitive, the measurement is time-consuming and measured values can vary considerably between laboratories(14). In aldosteronism with suppressed renin, the ratio of ARR is clearly dependent on the variants lower detection limit(15). Though determination of ARC in contrast to PRA offers advantage with regard to processing and standardization, knowing the postcaptopril sensitivity and specificity as well as the optimum cut off value of ARC is paramount (16) help to the diagnosis PA (15, 17, 18) and might serve better performance than ARRPRA.

ELIGIBILITY:
Inclusion Criteria:

1. age at onset younger than 35 years,
2. hypertension that is difficult to control after initiating therapy,
3. clinical occurrence of a hypertensive crisis,
4. the presence of hypokaliemia or metabolic alkalosis, or a random aldosterone-renin ration (ARR) >30, and
5. evidence of adrenal incidentaloma and hypertension or hypokalemia.

Exclusion Criteria:

1. chronic kidney disease with elevated estimated glomerular filtration rate (< 60, mL/min/1.73 m2)
2. liver disease with elevated GPT (> 35)
3. heart failure
4. classified as more than NYHA II,
5. hyperthyroidism
6. malignancy with metastasis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were referred to the hypertension clinics for suspicious of aldosteronism after an initial evaluation, and recorded in the Taiwan Primary Aldosteronism Investigation (TAIPAI). The initial evaluation included (1) age at onset younger than 35 years, (2) hypertension that is difficult to control after initiating therapy, (3) clinical occurrence of a hypertensive crisis, (4) the presence of hypokaliemia or metabolic alkalosis, or a random aldosterone-renin ration (ARR) >30, and (5) evidence of adrenal incidentaloma and hypertension or hypokalemia. All patients with intention to confirm and received captopril test were recruited and data were prospectively collected.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-01 (Estimated); Study Completion 2009-05 (Estimated)

PRIMARY OUTCOMES:
Determination of ARC in contrast to PRA offers advantage with regard to processing and standardization, knowing the postcaptopril sensitivity and specificity | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Sheu JY, Wang SM, Wu VC, Huang KH, Tseng CS, Lee YJ, Tsai YC, Lin YH, Chueh JS. Estimated glomerular filtration rate-dip after medical target therapy associated with increased mortality and cardiovascular events in patients with primary aldosteronism. J Hypertens. 2023 Sep 1;41(9):1401-1410. doi: 10.1097/HJH.0000000000003479. Epub 2023 Jun 8. PMID 37334546
- [Derived] Wu VC, Kuo CC, Chang HW, Tsai CT, Lin CY, Lin LY, Lin YH, Wang SM, Huang KH, Fang CC, Ho YL, Liu KL, Chang CC, Chueh SC, Lin SL, Yen RF, Wu KD; TAIPAI study group. Diagnosis of primary aldosteronism: comparison of post-captopril active renin concentration and plasma renin activity. Clin Chim Acta. 2010 May 2;411(9-10):657-63. doi: 10.1016/j.cca.2010.01.027. Epub 2010 Feb 1. PMID 20117105